CLINICAL TRIAL: NCT00836979
Title: Urinary Incontinence: Reproductive/Hormonal Risk Factors III
Brief Title: Urinary Incontinence: Reproductive/Hormonal Risk Factors
Acronym: RRISK3
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CN-08Svand-01-H; P50DK064538 (NIH)
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Incontinence; bladder problems; bladder dysfunction
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Sera will be banked for this cohort.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a continuation or follow-up of two previous studies (RRISK and RRISK2) conducted at the Kaiser Division of Research. This study will invite previous study participants, as well as a randomly selected group of Northern California Kaiser Permanente Members, to participate in an interview, mailed survey and lab visit. The purpose of this study is to examine the risk factors for bladder and pelvic problems.

DETAILED DESCRIPTION:
Using a cohort established during two previous studies (RRISK, CN-97Svand-01-H and RRISK2 CN-02Svand-07-H), this study will follow a well characterized cohort of middle-aged and older women who have been members of Kaiser Permanente Medical Care Plan (KPMCP) of Northern California continuously since age 18. The cohort is composed of over 2000 women for whom we have data from abstracted medical records, in-person interview, voiding diaries, physical assessments, laboratory data, and banked sera. Our cohort is unique in including a substantial number of women from the 4 major ethnic/race groups (white non-Hispanic, Black, Asian and Hispanic.) For this study, we will re-interview as many study participants from RRISK and RRISK2 as are willing. This study will also expand to further increase its diversity by adding a total of 450 Black, Asian and Hispanic women to the cohort. The overall goal of the study is to advance our understanding of mechanisms of Urinary Incontinence and facilitate the translational development of novel approaches to treatment and prevention.

ELIGIBILITY:
Inclusion Criteria:

* previously participated in the RRISK or RRISK2 studies at the kaiser Division of Research.

Exclusion Criteria:

* Not a part of the previous RRISK or RRISK2 cohorts.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A previously identified cohort of approximately 2000 women who are members of Kaiser Permanente Northern California (KPNC) health plan, having seen a Provider for bladder/incontinence related issues and have previously participated in the RRISK and RRISK2 studies. We will also randomly identify an additional cohort of women who are current members KPNC which report race/ethnicity as Asian, Hispanic or Black/African American (to total an additional 450 women across all groups.)
Sampling Method: Non-Probability Sample
Enrollment: 2161 (Actual)
Dates: Start 2008-10; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Race/Ethnicity | up to 48 months
  To investigate the two- to three-fold greater prevalence of stress UI in White women, compared to Black and Asian women which we previously reported we will (a) create and compare risk factor models of UI for each racial/ethnic group (White, Black, Hispanic, Asian); b) determine the extent to which racial differences can be explained by differences in newly measured exposures and genetic polymorphisms in addition to previously identified risk factors. To increase study power, we will enroll an additional 450 women (150 Black, 150 Asian and 150 Hispanic) into the RRRISK cohort.

OTHER OUTCOMES:
Hormones | up to 48 months
  To further characterize the association between hormones and UI and to determine if phytoestrogens are a risk factor for UI we will (a) use pharmacy records, supplemented by self-report, to ascertain the type, dose, duration and delivery for estrogens and for selective estrogen reuptake inhibitors (SERMs) and test their association with UI; (b) estimate phytoestrogen exposure from self-reported intake of key foods and botanicals and test the association with UI using multivariate analysis.
Gene Polymorphisms | up to 48 months
  To test the association between estrogen receptor gene polymorphisms and UI we will use banked serum samples from the RRISK cohort to assay for polymorphisms of the two estrogen receptor genes (ESR1 and ESR2) and determine their associations with urinary incontinence.
New UI and Progressive UI | up to 48 months
  We will analyze approximately 20,000 person-years of observational data using multiple regression techniques to (a) determine rates of new UI and changes in UI frequency/severity (including remission) and (b) identify risk factors for new UI and change in UI severity.
Pre-Diabetes | up to 48 months
  To investigate the association between pre-diabetes and increased risk of UI recently reported by members of our group we will (a) examine the cross-sectional association between pre-diabetes and UI, controlling for multiple other variables including body mass, waist circumference, inflammatory markers, and coronary heart disease; (b) conduct in-person interviews, measure physical parameters, and obtain blood tests on the approximately 400 women in the current study cohort with pre-diabetes. This additional prospective data on pre-diabetic women will allow us to characterize the natural history of the association between pre-diabetes and progression or new onset of UI.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen K Van Den Eeden, PhD, Principal Investigator — Kaiser Division of Research; Jeanette Brown, MD, Principal Investigator — UCSF/Mr. Zion WHCRC; David Thom, MD, Principal Investigator — UCSF/Family and Community Medicine
Locations (1):
- Kaiser Division of Research, Oakland, California, United States